CLINICAL TRIAL: NCT03644836
Title: Interest of Branched Chain Amino Acids Associated With a Respiratory Rehabilitation Program in Patients Broncho Chronic Obstructive Pulmonary Disease. Randomized Study Against Placebo
Brief Title: Interest of Branched Chain Amino Acids Associated With a Respiratory Rehabilitation Program in Patients Broncho Chronic Obstructive Pulmonary Disease
Acronym: REHABAAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REHABAAR
Record Dates: First submitted 2018-08-06; First posted 2018-08-23 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Broncho Chronic Obstructive Pulmonary Disease
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retraining with respiratory effort+ amino acids (Experimental)
  Interventions: Drug: Amino Acids
- Retraining with respiratory effort+ placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Amino Acids — Sweet taste cocoa flavored drink
  Arms: Retraining with respiratory effort+ amino acids
Drug: Placebos — Sweet taste cocoa flavored drink
  Arms: Retraining with respiratory effort+ placebo

SUMMARY:
Respiratory rehabilitation is one of the main treatments for COPD in the early stages of the disease (Stage 2 of GOLD) with a recognized effect on improving the capacity of the patients to exert effort by fighting against deconditioning. the effort. This treatment also improves the quality of life of patients and reduces the risk of respiratory exacerbations. The patients are very often malnourished and various studies have proposed the addition of oral supplementation such as hormone therapy (testosterone) to improve the exercise performance of these atrophied muscles. The use of branched-chain amino acids (AARs) such as valine, leucine, isoleucine in this indication can be fully justified because they stimulate protein synthesis and promote muscle maintenance and repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients Broncho Chronic Obstructive Pulmonary Disease in stages 2 and 3 of the GOLD classification, whose Maximum Expiratory Volume on the first second is between 30% and 80% of the expected theoretical value, associated with a maximal expiratory volume ratio on the first Second / Vital Capacity less than or equal to 70% of the expected theoretical value.
* Patients of both sexes, aged 40 to 80 years
* In case of active smoking, patients must commit to interrupting it during the respiratory rehabilitation program that will be proposed to them in this study

Exclusion Criteria:

* - Age <40 years or> 80 years
* Patients with a contraindication to exercise,
* Phenylketonuria
* Patients treated with long-term oxygen therapy and / or home ventilation will not be included.
* Patients with acute respiratory decompensation in the three months prior to inclusion.
* Patients with known allergy to milk, gluten, soy, egg and nuts
* Patients taking part in another clinical trial or who have participated in a clinical trial in the 3 months preceding this study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
maximum oxygene uptake | after 6 weeks of treatment
  maximum oxygene uptake measured during intensive exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude MEURICE, Principal Investigator — Poitiers University Hospital
Locations (1):
- Chu de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No